CLINICAL TRIAL: NCT00898716
Title: Phase 1 Multiple Ascending Dose Study of BMS-754807 in Patients With Solid Tumors in Japan
Brief Title: Multiple Ascending Dose Study of BMS-754807 in Patients With Solid Tumors in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA191-003
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2010-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BMS 754807

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-754807 (Experimental)
  Interventions: Drug: BMS-754807

INTERVENTIONS:
Drug: BMS-754807 — Tablets, Oral, 20 mg, 30 mg, 50 mg, 70 mg, 100 mg, 130 mg, 160 mg, 200 mg once daily, 3-5 months, depending on response

SUMMARY:
The purpose of this clinical study is to establish the maximum tolerated dose of BMS-754807 when administered orally on a once daily schedule in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group performance 0-1

Exclusion Criteria:

* Any disorder with dysregulation of glucose homeostasis
* Dumping syndrome
* History of glucose intolerance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose of BMS-754807 based on the Dose Limited Toxicity which observed during the first 28 days | Within the first 28 days

SECONDARY OUTCOMES:
To assess the safety and tolerability | Day 1, 8, 15, 22, 29, thereafter every 2 weeks
To establish recommended Phase 2 dose of BMS-754807 when administered orally on a once daily schedule | Day 1, 8, 15, 22, 29, thereafter every 2 weeks
To assess the metabolic effect on blood glucose | Day 1, 8, 15, 22, 29, thereafter every 2 weeks
To assess the pharmacokinetics of BMS-754807 administered orally on a once daily schedule | Day 1, 8, 15, 22, 29, thereafter every 2 weeks
To assess any preliminary evidence of anti-tumor activity | Day 1, 8, 15, 22, 29, thereafter every 2 weeks
To explore potential biomarkers of biological response | Day 1, 8, 15, 22, 29, thereafter every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-Ku, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx